CLINICAL TRIAL: NCT00614666
Title: Phase I/II Evaluation of the Safety, Pharmacokinetics, and Preliminary Effectiveness of Nikkomycin Z in the Treatment of Patients With Uncomplicated Coccidioides Pneumonia
Brief Title: Safety and PK of Nikkomycin Z for Coccidioides Pneumonia Treatment
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Recruitment challenges and lack of funding caused an early end to this study
Sponsor: University of Arizona (Other)
Collaborators: FDA Office of Orphan Products Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: VCFE-2007-001
Record Dates: First submitted 2008-01-31; First posted 2008-02-13 (Estimated); Results first posted 2025-04-16 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-01

CONDITIONS: Coccidioidomycosis
Keywords: coccidioidomycosis; Valley Fever; nikkomycin Z
MeSH Terms: conditions — Coccidioidomycosis | interventions — nikkomycin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- A - First dose level (n=5) (Experimental): nikkomycin Z 50 mg BID x 14 days
  Interventions: Drug: nikkomycin Z
- B - Second Dose Level (n=10) (Experimental): nikkomycin Z nikkomycin Z 250 mg BID x 14 days
  Interventions: Drug: nikkomycin Z
- C - Third Dose Level (n=10) (Experimental): nikkomycin Z 500 mg BID x 14 days
  Interventions: Drug: nikkomycin Z
- D - Fourth Dose Level (n=5) (Experimental): nikkomycin Z 750 BID x 14 days
  Interventions: Drug: nikkomycin Z
- Placebo (Placebo Comparator): placebo BID x 14 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: nikkomycin Z — Stage I: Multiple rising doses. Doses packaged on a unit dose basis in 50 and 250 mg capsules. Subjects take 1-3 capsules per dosing block for 14 days unless ADE or study withdrawal. Dose escalation unless a dose-limiting adverse effect is noted. Subjects assigned to BID dosing will receive 28 doses and subjects assigned to TID dosing will receive 42 doses.
  * 50 mg BID (n=4) vs placebo capsule BID (n=1)
  * 50 mg BID (n=4) vs 250 mg BID (n=4) vs Placebo capsule BID (n=2)
  * 250 mg BID (n=4) vs 500 mg BID (n=4) vs Placebo capsule BID (n=2)
  * 500 mg BID (n=4) vs Placebo capsule BID (n=1)
  At least 4 subjects complete lower dose before randomization includes next higher dose.
  Stage II will be a single dose level selected based on pharmacodynamics and safety from Stage I for 20 additional subjects using 4:1 randomization.
  Arms: A - First dose level (n=5); B - Second Dose Level (n=10); C - Third Dose Level (n=10); D - Fourth Dose Level (n=5)
Drug: Placebo — Placebo comparator
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine if nikkomycin Z is safe when administered at different dose levels for 14 days. The study will also determine blood levels and urinary excretion of nikkomycin Z in relation to dose administered. Patients with mild forms of Valley Fever pneumonia will be eligible to participate and will be allocated to receive treatment with nikkomycin Z (various doses) or a placebo. A secondary goal of this study is to evaluate the effectiveness and dose response of nikkomycin Z in an exploratory analysis.

DETAILED DESCRIPTION:
Every year there are 50,000 new U.S. cases of coccidioidomycosis (Valley Fever). The majority of these illnesses occur as a result of endemic exposure in Arizona and California. The benefits of antifungal therapy for uncomplicated disease are not currently established. Current therapies for serious and complicated forms of coccidioidomycosis are only partially effective and in themselves are unable to eradicate the fungus from sites of infection, commonly resulting in breakthrough infection and/or relapse. Nikkomycin Z is effective in the mouse model and results in improved microbiological response over fluconazole.

The goals of this study include: 1) Evaluating the safety and tolerance of nikkomycin Z following administration of multiple doses (50 mg Q 12 h to 750 mg Q 8 h) for two week and 2) Evaluating the pharmacokinetics of nikkomycin Z after single and multiple doses in relationship to dose. The study will include patients with uncomplicated Coccidioides pneumonia (mild illness) which will allow exploratory analysis of efficacy and dose response based on biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years and <= 50 years
* Male or Female (if female, must have a negative pregnancy test and agree to use an acceptable contraception method)
* Able to understand study and give written informed consent
* Have a respiratory illness with at least one of the following: Cough, chest pain dyspnea or tachypnea, sputum production, or fever/chills/night sweats
* Have a new or suspected new pulmonary infiltrate on Chest X-ray
* Have a positive coccidioidal serology by EIA or immunodiffusion

Exclusion Criteria:

* Patients under the age of 18 years or over 50 years
* Patients with a prior history of confirmed coccidioidal infection
* Laboratory diagnosis of another etiology for the inclusion-defining illness
* Inability to comprehend study and provide informed consent
* History of or current evidence of major organ disease
* Concomitant use of prednisone and other corticosteroids not permitted
* Concomitant immunosuppressive therapy is not permitted
* Concomitant antibacterial therapy is not permitted

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2007-09; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David E Nix, Pharm D, Principal Investigator — University of Arizona
Locations (1):
- Clinical & Translational Research Center - University of Arizona, Tucson, Arizona, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data may be shared for legitimate use to further nikkomycin Z development.
Supporting Information: Study Protocol, ICF
Time Frame: Study was terminated due to poor enrollment. Study report was not generated beyond safety data.
Access Criteria: Contact Valley fever Solutions - current license for development.

REFERENCES:
- See also: The Valley Fever Center for Excellence — http://www.vfce.arizona.edu

RESULTS

PARTICIPANT FLOW:
Groups:
- A - First Dose Level: nikkomycin Z 50 mg BID x 14 days
  nikkomycin Z: Stage I: Multiple rising doses. Doses packaged on a unit dose basis in 50 and 250 mg capsules. Subjects take 1-3 capsules per dosing block for 14 days unless ADE or study withdrawal. Dose escalation unless a dose-limiting adverse effect is noted. Subjects assigned to BID dosing will receive 28 doses and subjects assigned to TID dosing will receive 42 doses.
  * 50 mg BID vs placebo capsule BID
  * 50 mg BID vs 250 mg BID vs Placebo capsule BID
  * 250 mg BID vs 500 mg BID vs Placebo capsule BID
  * 500 mg BID vs Placebo capsule BID
  At least 4 subjects complete lower dose before randomization includes next higher dose.
  Stage II will be a single dose level selected based on pharmacodynamics and safety from Stage I for 20 additional subjects using 4:1 randomization.
- B - Second Dose Level: nikkomycin Z nikkomycin Z 250 mg BID x 14 days
  nikkomycin Z: Stage I: Multiple rising doses. Doses packaged on a unit dose basis in 50 and 250 mg capsules. Subjects take 1-3 capsules per dosing block for 14 days unless ADE or study withdrawal. Dose escalation unless a dose-limiting adverse effect is noted. Subjects assigned to BID dosing will receive 28 doses and subjects assigned to TID dosing will receive 42 doses.
  * 50 mg BID vs placebo capsule BID
  * 50 mg BID vs 250 mg BID vs Placebo capsule BID
  * 250 mg BID vs 500 mg BID vs Placebo capsule BID
  * 500 mg BID vs Placebo capsule BID
  At least 4 subjects complete lower dose before randomization includes next higher dose.
  Stage II will be a single dose level selected based on pharmacodynamics and safety from Stage I for 20 additional subjects using 4:1 randomization.
- C - Third Dose Level: nikkomycin Z 500 mg BID x 14 days
  nikkomycin Z: Stage I: Multiple rising doses. Doses packaged on a unit dose basis in 50 and 250 mg capsules. Subjects take 1-3 capsules per dosing block for 14 days unless ADE or study withdrawal. Dose escalation unless a dose-limiting adverse effect is noted. Subjects assigned to BID dosing will receive 28 doses and subjects assigned to TID dosing will receive 42 doses.
  * 50 mg BID vs placebo capsule BID
  * 50 mg BID vs 250 mg BID vs Placebo capsule BID
  * 250 mg BID vs 500 mg BID vs Placebo capsule BID
  * 500 mg BID vs Placebo capsule BID
  At least 4 subjects complete lower dose before randomization includes next higher dose.
  Stage II will be a single dose level selected based on pharmacodynamics and safety from Stage I for 20 additional subjects using 4:1 randomization.
- D - Fourth Dose Level: nikkomycin Z 750 BID x 14 days
  nikkomycin Z: Stage I: Multiple rising doses. Doses packaged on a unit dose basis in 50 and 250 mg capsules. Subjects take 1-3 capsules per dosing block for 14 days unless ADE or study withdrawal. Dose escalation unless a dose-limiting adverse effect is noted. Subjects assigned to BID dosing will receive 28 doses and subjects assigned to TID dosing will receive 42 doses.
  * 50 mg BID vs placebo capsule BID
  * 50 mg BID vs 250 mg BID vs Placebo capsule BID
  * 250 mg BID vs 500 mg BID vs Placebo capsule BID
  * 500 mg BID vs Placebo capsule BID
  At least 4 subjects complete lower dose before randomization includes next higher dose.
  Stage II will be a single dose level selected based on pharmacodynamics and safety from Stage I for 20 additional subjects using 4:1 randomization.
Period: Overall Study
Arm/Group | A - First Dose Level | B - Second Dose Level | C - Third Dose Level | D - Fourth Dose Level | Placebo
Started | 4 | 1 | 0 | 0 | 1
Completed | 4 | 1 | 0 | 0 | 1
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- A - First Dose Level (n=5): nikkomycin Z 50 mg BID x 14 days
  nikkomycin Z: Stage I: Multiple rising doses. Doses packaged on a unit dose basis in 50 and 250 mg capsules. Subjects take 1-3 capsules per dosing block for 14 days unless ADE or study withdrawal. Dose escalation unless a dose-limiting adverse effect is noted. Subjects assigned to BID dosing will receive 28 doses and subjects assigned to TID dosing will receive 42 doses.
  * 50 mg BID (n=4) vs placebo capsule BID (n=1)
  * 50 mg BID (n=4) vs 250 mg BID (n=4) vs Placebo capsule BID (n=2)
  * 250 mg BID (n=4) vs 500 mg BID (n=4) vs Placebo capsule BID (n=2)
  * 500 mg BID (n=4) vs Placebo capsule BID (n=1)
  At least 4 subjects complete lower dose before randomization includes next higher dose.
  Stage II will be a single dose level selected based on pharmacodynamics and safety from Stage I for 20 additional subjects using 4:1 randomization.
- B - Second Dose Level (n=10): nikkomycin Z nikkomycin Z 250 mg BID x 14 days
  nikkomycin Z: Stage I: Multiple rising doses. Doses packaged on a unit dose basis in 50 and 250 mg capsules. Subjects take 1-3 capsules per dosing block for 14 days unless ADE or study withdrawal. Dose escalation unless a dose-limiting adverse effect is noted. Subjects assigned to BID dosing will receive 28 doses and subjects assigned to TID dosing will receive 42 doses.
  * 50 mg BID (n=4) vs placebo capsule BID (n=1)
  * 50 mg BID (n=4) vs 250 mg BID (n=4) vs Placebo capsule BID (n=2)
  * 250 mg BID (n=4) vs 500 mg BID (n=4) vs Placebo capsule BID (n=2)
  * 500 mg BID (n=4) vs Placebo capsule BID (n=1)
  At least 4 subjects complete lower dose before randomization includes next higher dose.
  Stage II will be a single dose level selected based on pharmacodynamics and safety from Stage I for 20 additional subjects using 4:1 randomization.
- C - Third Dose Level (n=10): nikkomycin Z 500 mg BID x 14 days
  nikkomycin Z: Stage I: Multiple rising doses. Doses packaged on a unit dose basis in 50 and 250 mg capsules. Subjects take 1-3 capsules per dosing block for 14 days unless ADE or study withdrawal. Dose escalation unless a dose-limiting adverse effect is noted. Subjects assigned to BID dosing will receive 28 doses and subjects assigned to TID dosing will receive 42 doses.
  * 50 mg BID (n=4) vs placebo capsule BID (n=1)
  * 50 mg BID (n=4) vs 250 mg BID (n=4) vs Placebo capsule BID (n=2)
  * 250 mg BID (n=4) vs 500 mg BID (n=4) vs Placebo capsule BID (n=2)
  * 500 mg BID (n=4) vs Placebo capsule BID (n=1)
  At least 4 subjects complete lower dose before randomization includes next higher dose.
  Stage II will be a single dose level selected based on pharmacodynamics and safety from Stage I for 20 additional subjects using 4:1 randomization.
- D - Fourth Dose Level (n=5): nikkomycin Z 750 BID x 14 days
  nikkomycin Z: Stage I: Multiple rising doses. Doses packaged on a unit dose basis in 50 and 250 mg capsules. Subjects take 1-3 capsules per dosing block for 14 days unless ADE or study withdrawal. Dose escalation unless a dose-limiting adverse effect is noted. Subjects assigned to BID dosing will receive 28 doses and subjects assigned to TID dosing will receive 42 doses.
  * 50 mg BID (n=4) vs placebo capsule BID (n=1)
  * 50 mg BID (n=4) vs 250 mg BID (n=4) vs Placebo capsule BID (n=2)
  * 250 mg BID (n=4) vs 500 mg BID (n=4) vs Placebo capsule BID (n=2)
  * 500 mg BID (n=4) vs Placebo capsule BID (n=1)
  At least 4 subjects complete lower dose before randomization includes next higher dose.
  Stage II will be a single dose level selected based on pharmacodynamics and safety from Stage I for 20 additional subjects using 4:1 randomization.
- Total: Total of all reporting groups
Arm/Group | A - First Dose Level (n=5) | B - Second Dose Level (n=10) | C - Third Dose Level (n=10) | D - Fourth Dose Level (n=5) | Placebo | Total
Number analyzed (Participants) | 4 | 1 | 0 | 0 | 1 | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 4 | 1 | 0 | 0 | 1 | 6
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 0 | 0 | 1 | 2
  Male | 3 | 1 | 0 | 0 | 0 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 4 | 1 | 0 | 0 | 1 | 6
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0
  White | 4 | 1 | 0 | 0 | 1 | 6
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 4 | 1 |  |  | 1 | 6

OUTCOME MEASURES:

1. Primary Outcome: Concentration of Nikkomycin Z in the Blood Over Time (AUC)
Time Frame: 0, 0.25, 0.5, 0.75, 1.0, 1.5, 2 , 3, 4, 6, 8 and 12 h hours post-dose on Day 1 and Day 14
Population: The study was terminated after enrollment of 6 subjects
Measure: Mean (Standard Deviation); unit: mg*hr/L
Arm/Group | A - First Dose Level (n=5) | B - Second Dose Level (n=10) | C - Third Dose Level (n=10) | D - Fourth Dose Level (n=5)
Number analyzed (Participants) | 4 | 1 | 0 | 0
mg*hr/L
  Day 1 | 3.444 (0.710) | 19.923 (NA) — Standard Deviation not calculable for 1 participant |  |
  Day 14 | 3.900 (1.583) | 24.045 (NA) — Standard Deviation not calculable for 1 participant |  |

2. Primary Outcome: Highest Concentration of Nikkomycin Z in the Blood (Cmax)
Time Frame: 0, 0.25, 0.5, 0.75, 1.0, 1.5, 2 , 3, 4, 6, 8 and 12 h hours post-dose on Day 1 and Day 14
Population: The study was terminated after enrollment of 6 subjects
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | A - First Dose Level (n=5) | B - Second Dose Level (n=10) | C - Third Dose Level (n=10) | D - Fourth Dose Level (n=5)
Number analyzed (Participants) | 4 | 1 | 0 | 0
mg/L
  Day 1 | 0.710 (0.188) | 3.748 (NA) — Standard Deviation not calculable for 1 participant |  |
  Day 14 | 0.811 (0.248) | 4.275 (NA) — Standard Deviation not calculable for 1 participant |  |

ADVERSE EVENTS:
Arm/Group | A - First Dose Level (n=5) | B - Second Dose Level (n=10) | C - Third Dose Level (n=10) | D - Fourth Dose Level (n=5) | Placebo
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/1 | 0/0 | 0/0 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/1 | 0/0 | 0/0 | 0/1
Other Adverse Events (participants affected / at risk) | 3/4 | 1/1 | 0/0 | 0/0 | 1/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | A - First Dose Level (n=5) (N=4) | B - Second Dose Level (n=10) (N=1) | C - Third Dose Level (n=10) (N=0) | D - Fourth Dose Level (n=5) (N=0) | Placebo (N=1)
Hypotension (Vascular disorders) | 1 (1) | 0 | 0 | 0 | 0
Near syncope (General disorders) | 1 (1) | 0 | 0 | 0 | 0
Headache (General disorders) | 3 (6) | 1 (1) | 0 | 0 | 1 (5)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 | 0 | 0 | 0
Dry mouth (General disorders) | 1 (1) | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 (1) | 0 | 0 | 0 | 1 (1)
Insomnia (General disorders) | 1 (1) | 0 | 0 | 0 | 0
Cataract surgery (Eye disorders) | 1 (1) | 0 | 0 | 0 | 0
Left lung nodule (Respiratory, thoracic and mediastinal disorders) | 0 | 1 (1) | 0 | 0 | 0
Right temple pain (General disorders) | 0 | 1 (1) | 0 | 0 | 0

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of subjects analyzed

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes